CLINICAL TRIAL: NCT01317069
Title: A Randomized, Open, Prospective Clinical Research Programs of Fluorouracil Implant (Sinofuan) to Improve Surgical Gallbladder Cancer and Bile Duct Cancer
Brief Title: A Randomized, Open, Prospective Clinical Research of Fluorouracil Implant to Improve Surgical Gallbladder Cancer and Bile Duct Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Simcere Pharmaceutical Co., Ltd (Other)
Collaborators: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Yongjie Zhang MD, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sinofuan201101
Record Dates: First submitted 2011-03-15; First posted 2011-03-17 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Gallbladder Cancer; Bile Duct Cancer
MeSH Terms: conditions — Gallbladder Neoplasms; Bile Duct Neoplasms | interventions — Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fluorouracil implant (Experimental)
  Interventions: Drug: Fluorouracil implant

INTERVENTIONS:
Drug: Fluorouracil implant — Before the abdomen was closed, fluorouracil implant 1000mg was sprayed evenly on the surface of tumor resection area, and some of the drugs were put into mesenteric root based on the location
  Other Names: Sinofuan

SUMMARY:
Through clinical practice, to explore if the application of Fluorouracil implant could effectively delay the local tumor recurrence and improvement the postoperative survival time in patients with gallbladder cancer and bile duct cancer.

DETAILED DESCRIPTION:
Major Objective Through clinical practice, to explore if the application of Fluorouracil implant could effectively delay the local tumor recurrence and improvement the postoperative survival time in patients with gallbladder cancer and bile duct cancer.

Secondary objective

1) If Fluorouracil implants application in clinical surgery could lead to the incidence of complications increased in biliary-enteric anastomosis.

2）Assess drug safety according to drug-related clinical and / or laboratory adverse events.

3）Observe the postoperative complication rate of Fluorouracil implants. 4）Observe the quality of life of patients used Fluorouracil implants.

ELIGIBILITY:
Inclusion Criteria:

* The patients with gallbladder and bile duct cancer diagnosis by surgical exploration, or intraoperative frozen biopsy (Annex 2).
* Aged 18 to 70 years old, male or female, body condition score generally ECOG 0～2, expected survival ≥ 3 months.
* Subjects were no major organ dysfunction, blood, liver, kidney and heart function was normal, the specific requirements of laboratory indicators:

Blood: WBC count > 3.0 × 109 / L, Platelet count> 100 × 109 / L, Hb > 8.0g/dl. Liver function：serum bilirubin less than 1.5 times the upper limit of normal; ALT and AST less than 3 times the upper limit of normal.

Renal function: creatinine less than 1.5 times the upper limit of normal.

* Participants have used other chemotherapy drugs, subject to the 30-day washout period before proceeding with the test.
* Patients had no anaphylactic reaction with oxaliplatin and fluorouracil in the past.
* Patients who can understand the circumstances of this study and signed informed consent.

Exclusion Criteria:

* Currently is receiving effective treatment；
* Pregnancy, breast-feeding patients；
* Primary brain tumors or central nervous system metastatic tumor is not controlled;
* Patients received chemotherapy, radiotherapy, biological therapy, other drugs or instrument therapy 30 days before enrollment.
* Patients with purulent and chronic infected wounds which delayed healing.
* Patients with liver, kidney and heart failure and coronary heart disease, angina, myocardial infarction, arrhythmia, cerebral thrombosis, stroke and other serious cardiovascular and cerebrovascular disease;
* Patients has a history of mental illness and difficult to control;
* Patients who was considered inappropriate to participate in the trials by the researchers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-12 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
duration of survival after operation | 3 years

SECONDARY OUTCOMES:
disease free survival | 1 years

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality, China